CLINICAL TRIAL: NCT06886659
Title: A Randomized, Double Blind, Parallel, Active Controlled Study to Compare PK, Immunogenicity and Safety of Trastuzumab of Incepta With Trastuzumab (Roche) in Healthy, Adult Subjects by Single IV Infusion Under Fasting Condition
Brief Title: A Study to Compare PK, Immunogenicity and Safety of Trastuzumab of Incepta Pharmaceuticals Ltd With Trastuzumab (Roche)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incepta Pharmaceuticals Ltd (Industry)
Collaborators: EskeGen Ltd, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/TR/P-I/01
Record Dates: First submitted 2025-01-12; First posted 2025-03-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Disease; Antineoplastic Agents
Keywords: Biosimilarity; Bioequivalence; Tastuzumab; Healthy male volunteers; PK
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial. Assignment to a group will be randomized.
Who Masked: Participant, Investigator
Masking Description: Subjects will be administered either the Test or Reference product, according to the randomization schedule. The test and reference product will be assigned with the randomization code A and B respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trastuzumab (proposed Trastuzumab biosimilar) (Experimental): 40 healthy adult male will get Trastuzumab 150 mg/vial manufactured by Incepta Pharmaceuticals Ltd.
  Interventions: Drug: Trastuzumab (proposed Trastuzumab biosimilar)
- Herclon (Active Comparator): 40 healthy adult male will get Herclon 150 mg/vial manufactured by Roche.
  Interventions: Drug: Herclon

INTERVENTIONS:
Drug: Trastuzumab (proposed Trastuzumab biosimilar) — 6 mg/kg single intravenous infusion of Trastuzumab of Incepta Pharmaceuticals Ltd
  Other Names: Test Product
  Arms: Trastuzumab (proposed Trastuzumab biosimilar)
Drug: Herclon — 6 mg/kg single intravenous infusion of Trastuzumab of Roche
  Other Names: Reference Product
  Arms: Herclon

SUMMARY:
Trastuzumab is an Ig G1 kappa, humanized monoclonal antibody which is most abundant subclass of IgG, that works against overexpress of HER2 (Human Epidermal Growth Factor Receptor Type 2). Trastuzumab is used to treat HER2-positive breast, gastroesophageal, and gastric cancers. HER2 regulate cell growth and survival, as well as adhesion, migration, differentiation and other cellular response. But when HER2 signaling is over expressed it causes uncontrolled cell growth which leads to the formation of cancerous tumor.

DETAILED DESCRIPTION:
In this study, healthy adult male volunteers will receive a single intravenous administration of Trastuzumab (Incepta) or Trastuzumab (Roche) according to randomization. During the course of the study, the pharmacokinetics will be assessed by sampling the levels of the drug in the blood and by comparing these levels among the different administration arms. Safety and immunologic response will also be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male participant, age 18 to 55 years old
* BMI 18.5 to 30.0 weight in kg/height in meter2; BMI value should be rounded off to one significant digit after decimal point. Volunteer having body weight at least 50 Kg.
* Non-smokers and non-tobacco user (i.e. having no past history of smoking and tobacco consuming for at least one year prior to study)
* Able to understand procedure, agree to participate and willing to give informed consent.
* Willing and able to comply with the study procedures, restrictions and requirements as judged and confirmed by the principal investigator
* Male subjects, if married, must agree that they and their spouse will use adequate contraception or be of non-childbearing potential.

Exclusion Criteria:

* Have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination, vital signs, laboratory evaluations, ECG, Echocardiography (LVEF less than 55%)]. Any disease or condition like diabetes, psychosis or others which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, ophthalmic, pulmonary, metabolic, endocrine, immunological, respiratory, central nervous system or any other body system.
* History of and/or current cardiac disease
* Neutrophil count less than the lower limit of normal range during screening.
* A positive hepatitis screen (includes subtypes B & C).
* Use of hematopoietic growth factors, monoclonal antibodies or immunoglobulins within last 6 months prior to the study medication administration.
* History of any cancer, including carcinoma in situ
* Volunteer with history of angina, dyspnea, orthopnea, congestive heart failure or myocardial infarction
* Have received live vaccine(s) within 30 days prior to Screening or who will require a vaccine(s) between Screening and the End of Study visit.
* History or evidence of drug abuse or of alcoholism or of moderate alcohol use.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only adult male subjects will be enrolled for the study
Enrollment: 80 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Cmax | 71 days from the starting of infusion
  Maximum Observed Drug Concentration In Plasma
AUC0-t | 71 days from the starting of infusion
  Area Under The Concentration Versus Time Curve Up To The Last Measurable Time Point
AUC0-inf | 71 days from the starting of infusion
  Area Under The Concentration Versus Time Curve From Time 0 To Infinity
Safety assessment: The number of adverse events will be evaluated and compared between the reference and test drugs groups. | 71 days from the starting of infusion
  No of adverse events in both reference and test product arm will be assessed and compared by monitoring the presence of any AEs or SAEs throughout the study period.
Immunogenicity assessment: Immunogenicity will be assessed by measuring Anti-Drug Antibodies (ADA) formation. | 71 days from the starting of infusion
  The incidence of Anti-Drug Antibodies (ADA) formation will be measured by taking blood samples on before treatment (pre-dose) and and on day 71

CONTACTS AND LOCATIONS:
Overall Officials: Manindranath Roy, Principal Investigator — Professor (Biochemistry) United Medical College
Locations (2):
- Bangladesh (2):
  - Al-Manar Hospital Ltd,, Dhaka
  - Universal Medical College, Dhaka

IPD SHARING:
Plan to Share IPD: Yes
By publication in the journal
Supporting Information: Study Protocol, CSR
Time Frame: After completion of study
Access Criteria: Journal